CLINICAL TRIAL: NCT00356980
Title: A Phase I Trial of TNF-Bound Colloidal Gold (CYT-6091) by Intravenous Administration in Subjects With Advanced Solid Organ Malignancies
Brief Title: TNF-Bound Colloidal Gold in Treating Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 060167; 06-C-0167; NCI-P6062; CYT-6091-06-01; CDR0000486917; NCT00328406 (obsolete NCT alias)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2012-03-15 (Estimated); Status verified 2012-03

CONDITIONS: Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific
MeSH Terms: interventions — CYT-6091

INTERVENTIONS:
Biological: colloidal gold-bound tumor necrosis factor
Other: pharmacological study

SUMMARY:
RATIONALE: Biological therapies, such as TNF-bound colloidal gold, may stimulate the immune system in different ways and stop tumor cells from growing.

PURPOSE: This phase I trial is studying the side effects and best dose of TNF-bound colloidal gold in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the maximum tolerated dose of TNF-bound colloidal gold (CYT-6091) in patients with advanced solid tumors.
* Determine the toxicities of CYT-6091 in these patients.

Secondary

* Determine the pharmacokinetics of CYT-6091 in these patients.
* Evaluate biopsy samples of tumor and adjoining normal tissue for levels of CYT-6091.
* Determine if antitumor effects of CYT-6091 occur in these patients.

OUTLINE: This is an open-label, sequential cohort, dose-escalation study.

Patients receive TNF-bound colloidal gold (CYT-6091) IV on days 1 and 15 (course 1). Approximately 4-6 weeks later, patients are re-staged and responding patients may receive another course of therapy. Patients may receive up to 3 re-treatment courses.

Cohorts of 3-6 patients receive escalating doses of CYT-6091 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 1 of 6 patients experience dose-limiting toxicity.

Blood samples are collected at baseline and periodically during the first course of therapy for pharmacokinetic and pharmacodynamic analyses.

After completion of study treatment, patients are followed every 3 months for 1 year, every 4 months for the next year, and then every 6 months thereafter.

PROJECTED ACCRUAL: A total of 60 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed solid tumor
* Advanced and/or metastatic disease
* Unresponsive to conventional therapy (i.e., disease progressed while receiving any known standard curative or palliative therapy) OR previously untreated tumor for which no standard treatment exists
* Measurable or evaluable metastatic disease
* No lymphoma or other hematologic malignancy
* No known brain metastases

  * Previously treated brain metastases with no evidence of recurrence allowed

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Life expectancy ≥ 3 months
* Absolute neutrophil count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* Creatinine ≤ 2.0 mg/dL
* Bilirubin ≤ 2.5 mg/dL
* ALT and AST ≤ 1.5 times upper limit of normal (ULN) (3 times ULN if liver metastases are present)
* Alkaline phosphatase ≤ 1.5 times ULN (3 times ULN if liver metastases are present)
* Prothrombin time ≤ 1.5 times ULN
* Hemoglobin ≥ 10.0 g/dL (transfusion allowed)
* LVEF ≥ 45% by echocardiogram or thallium stress test for patients > 50 years of age or history of cardiovascular disease
* FEV_1 and DLCO > 30% of predicted for patients with a history of pulmonary disease
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active bacterial or viral infection with systemic manifestations (e.g., fever, symptoms, leukocytosis)

  * Localized chronic infections, such as mild acne or tinea pedis allowed
* No acute or chronic viral hepatitis
* No known bleeding disorder
* No other concurrent life-threatening illness, including any of the following:

  * Unstable angina
  * Severe oxygen-dependent chronic obstructive pulmonary disease
  * End-stage liver disease
* No known active renal disease or renal insufficiency as evidenced by serum creatinine > 2.0 mg/dL
* No HIV positivity

PRIOR CONCURRENT THERAPY:

* Recovered from prior therapy
* More than 3 weeks since prior biological or cytotoxic agents (6 weeks for nitrosoureas)
* No known requirment for palliative treatment
* No concurrent surgery
* No other concurrent anticancer therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-02 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of TNF-bound colloidal gold (CYT-6091)
Toxicity

SECONDARY OUTCOMES:
Pharmacokinetic profile of CYT-6091
Measurements of CYT-6091 in tumor biopsies
Tumor biopsy histology and gene expression after treatment
Immunogenicity of CYT-6091
Electron microscopy of biopsy to determine presence of colloidal gold
Response of target and nontarget lesions
Overall response
Duration of response
Duration of stable disease

CONTACTS AND LOCATIONS:
Overall Officials: Steven K. Libutti, MD, Principal Investigator — NCI - Surgery Branch
Locations (2):
- United States (2):
  - Warren Grant Magnuson Clinical Center - NCI Clinical Trials Referral Office, Bethesda, Maryland
  - NCI - Surgery Branch, Bethesda, Maryland

REFERENCES:
- [Result] Libutti SK, Paciotti GF, Byrnes AA, Alexander HR Jr, Gannon WE, Walker M, Seidel GD, Yuldasheva N, Tamarkin L. Phase I and pharmacokinetic studies of CYT-6091, a novel PEGylated colloidal gold-rhTNF nanomedicine. Clin Cancer Res. 2010 Dec 15;16(24):6139-49. doi: 10.1158/1078-0432.CCR-10-0978. Epub 2010 Sep 27. PMID 20876255
- [Derived] Kesharwani P, Ma R, Sang L, Fatima M, Sheikh A, Abourehab MAS, Gupta N, Chen ZS, Zhou Y. Gold nanoparticles and gold nanorods in the landscape of cancer therapy. Mol Cancer. 2023 Jun 21;22(1):98. doi: 10.1186/s12943-023-01798-8. PMID 37344887